CLINICAL TRIAL: NCT03297450
Title: The Neuromodulatory Effect of Combined Transcranial Direct Current Stimulation (tDCS) with Aphasia Therapy in the Acute Phase After Ischemic Stroke
Brief Title: TDCS and Aphasia Therapy in the Acute Phase After Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult patient recruitment
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC2017/0906
Record Dates: First submitted 2017-09-05; First posted 2017-09-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-01

CONDITIONS: Aphasia Following Cerebral Infarction
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: aphasia therapy (45 minutes) in combination with (sham or real) tDCS (20 minutes)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Aphasia therapy and tDCS (Active Comparator)
  Interventions: Device: tDCS; Behavioral: Aphasia therapy
- Aphasia therapy and sham-tDCS (Sham Comparator)
  Interventions: Behavioral: Aphasia therapy; Device: Sham-tDCS
- Standard of care and sham-tDCS (Sham Comparator)
  Interventions: Device: Sham-tDCS

INTERVENTIONS:
Device: tDCS — C-tDCS during the first 20 minutes of aphasia therapy, at an intensity of 1mA
  Arms: Aphasia therapy and tDCS
Behavioral: Aphasia therapy — Based on linguistic tests, individualized aphasia therapy will be provided
  Arms: Aphasia therapy and sham-tDCS; Aphasia therapy and tDCS
Device: Sham-tDCS — tDCS during the first 20 minutes of aphasia therapy at an intensity of 0mA (Sham)
  Arms: Aphasia therapy and sham-tDCS; Standard of care and sham-tDCS

SUMMARY:
This study evaluates the neuromodulatory effect of combined tDCS and aphasia therapy in patients in the acute stage after stroke. Half of the participants will receive aphasia therapy and tDCS, the other half will receive aphasia therapy and sham-tDCS.

DETAILED DESCRIPTION:
Aphasia is present in about one third of all stroke patients in the acute phase. The first few months after stroke, considerable spontaneous recovery is initiated, including neuronal plasticity and reorganization processes. Language recovery in aphasic stroke patients involves reorganization of brain functions. Longitudinal fMRI studies reveal that the right hemisphere shows increased activity at different times in the recovery process, but in the long-term is correlated with poorer performance. Left re-lateralization, if possible, seems to be the most effective in restoring language function. For a large subgroup of patients, aphasia therapy is not sufficient to resolve language deficits and not all patients are capable to endure intensive aphasia therapy. Therefore, non-invasive techniques (NIBS) such as transcranial direct current stimulation (tDCS) are currently explored as an add-on treatment to improve or accelerate therapy outcomes. tDCS is a painless and safe stimulation tool that modulates cortical excitability through weak polarizing currents (1 mA - 2 mA) between two electrodes. These weak currents are thought to induce a subthreshold shift of resting membrane potentials towards depolarization or hyperpolarization. The effects of stimulation depend on the polarity of the applied current relative to the axonal orientation. It has been found that tDCS not only triggers immediate aftereffects, but also long-lasting effects that persist beyond the stimulation time, even for up to 12 months. It was suggested that long-term potentiation (LTP) and long-term depression (LTD) might be responsible for these long-term effects, however the precise physiologic mechanisms of action are not yet fully understood.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with mild-moderate aphasia (Token Test Score between 7 and 40)
* Inclusion in the first few days after stroke (acute phase)
* Age 18 - 85 years
* Being right-handed
* Mothertongue: Dutch
* Able to undergo functional and specific linguistic testing and therapy in the acute phase following stroke
* Imaging (CT or MRI) prior to inclusion (standard of care)
* Signed Informed Consent

Exclusion Criteria:

* History of other diseases of the central nervous system, psychological disorders and (developmental) speech and or language disorders
* Serious non-linguistic, cognitive disorders (as documented in the patients' medical history and inquired in anamneses)
* Prior brain surgery
* Excessive use of alcohol or drugs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Change in naming performance | baseline, 1 week, 3 months, 6 months
  Naming performance will be assessed with the Boston Naming Test at baseline, immediately following therapy, and after 3 and 6 months
Change in Vital Parameters | baseline, 1 hour (each session)
  Blood pressure and heart rate will be measured before and after each session of treatment

SECONDARY OUTCOMES:
Change in tolerability (Visual analogue scale) | baseline, 1 hour (each session)
  A Visual analogue scale will assess tolerability before and immediately after each session
Change in Spontaneous Speech | baseline, 1 week, 3 months, 6 months
  A Semi-standardized interview of the AAT will assess functional communication at baseline, immediately after therapy, and at 3 and 6 months
Change in ERPs | baseline, 1 week, 3 months, 6 months
  Evoked potentials will be measured at baseline, immediately after treatment and after 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Veerle De Herdt, Prof. Dr., Principal Investigator — University Ghent
Locations (1):
- University Hospital Ghent, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No